CLINICAL TRIAL: NCT05513612
Title: Safety and Efficacy Study of Novel CAR-T Cell Therapy in the Treatment of Hematopoietic and Lymphoid Malignancies
Brief Title: Novel CAR-T Cell Therapy in the Treatment of Hematopoietic and Lymphoid Malignancies
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The study is not initiated and we want it to be withdrawn.
Sponsor: Shanghai Pudong Hospital (Other)
Collaborators: UTC Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-IIT-002-E03
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Acute Myeloid Leukemia (AML); B-cell Non-Hodgkin's Lymphoma (B-NHL); Multiple Myeloma (MM); T-Cell Leukemia/Lymphoma, Adult; B-cell Acute Lymphoblastic Leukemia (B-ALL)
Keywords: CD123 CAR-T; CD19 CAR-T; BCMA CAR-T; CD7 CAR-T; Hematopoietic and Lymphoid Malignancies
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Lymphoma, B-Cell; Multiple Myeloma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous CAR-T cells (Experimental): A conditioning chemotherapy regimen of fludarabine and cyclophosphamide will be administered followed by investigational treatment, CAR-T cells. CAR-T cells targeted CD19/BCMA/CD123/CD7 are autologous genetically modified T cells.
  Interventions: Biological: Autologous CAR-T cells; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: Autologous CAR-T cells — CAR-T cells will be infused intravenously.
Drug: Fludarabine — Administered according to package insert
  Other Names: Fludara
Drug: Cyclophosphamide — Administered according to package insert
  Other Names: Cytoxan

SUMMARY:
The primary purpose of this study is to determine the safety and efficacy of novel autologous CAR-T cells in patients with hematopoietic and lymphoid malignancies.

DETAILED DESCRIPTION:
Chimeric antigen receptor (CAR)-modified T cells targeted CD19 have demonstrated unprecedented successes. Besides CD19, many other molecules such as CD123, BCMA, and CD7 may be potential in developing the corresponding CAR-T cells to treat patients with hematopoietic and lymphoid malignancies. UTC Therapeutics Inc. have developed an efficient platform for constructing CAR-T cells that can remodel of tumor microenvironment and enhance the anti-tumor immune response and persistence of CAR-T cells. In this study, all eligible subjects will receive a conditioning chemotherapy regimen of fludarabine and cyclophosphamide followed by investigational treatment, CAR-T cells. Safety, efficacy, pharmacokinetic, and pharmacodynamic of the CAR-T cells will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and the willingness to sign informed consent.
2. Patients with relapsed or refractory Acute Myeloid Leukemia (AML), B-cell Non-Hodgkin's Lymphoma (B-NHL), Multiple Myeloma (MM), Adult T-cell Leukemia/Lymphoma (ATL), B-cell Acute Lymphoblastic Leukemia (B-ALL) after at least two cycles of first-line therapy or autologous hematopoietic stem cell transplantation (auto-HSCT).
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0~2.
4. Adequate organ functions:

   * Sufficient bone marrow function evaluated by investigator to receive lymphodepleting preparative regimen;
   * Serum creatinine (Cr) ≤ 1.5 × upper limit of normal (ULN), or creatinine clearance rate (as estimated by Cockcroft Gault) > 30 mL/min/1.73 m^2;
   * Alanine aminotransferase (ALT) ≤ 5×ULN; and total bilirubin (TBIL) <2.0mg/dL; TBIL of patients with Gilbert's Syndrome or liver involvement must less than 3.0 mg/dL;
   * Left ventricular ejection fraction (LVEF) > 40%.
5. Subjects who have previously received CD19 targeted therapy must have biopsy-proven lymphoma lesions still express CD19 antigen.

Exclusion Criteria:

1. Lymphomas involving only the central nervous system (CNS) (subjects with secondary CNS lymphomas are admitted).
2. History of another malignancy that has not been in remission for at least 2 year (the following conditions may be excluded from the 2-year restriction: non-melanoma skin cancer, completely resected stage I tumor with low probability of recurrence, limited-stage prostate cancer after treatment, biopsy-proven cervical carcinoma in situ, or PAP smear showing squamous epithelium internal lesions).
3. History of treatment with Alemtuzumab within 6 months prior to leukapheresis, or Fludarabine or Cladribine within 3 months prior to leukapheresis.
4. Active hepatitis C (HCV), hepatitis B (HBV), human immunodeficiency virus (HIV), or syphilis infection.
5. Uncontrolled fungal, bacterial, viral, or other infection.
6. Acute or chronic graft-versus-host disease (GVHD).
7. History of any of the following cardiovascular diseases within the past 6 months: Class III or IV heart failure as defined by the New York Heart Association (NYHA), cardiac angioplasty or stent, myocardial infarction, unstable angina, or other clinically significant heart disease.
8. History or clinical evidence of CNS disease.
9. Female subjects who are pregnant or lactating.
10. Prior CAR-T therapy or other genetically modified T cell therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
TEAEs | 4 weeks
  Incidence and severity of Treatment Emergent Adverse Event.
TRAEs | 4 weeks
  Incidence and severity of Treatment Related Adverse Events.
AESIs | 4 weeks
  Incidence and severity of AEs of Special Interest.

SECONDARY OUTCOMES:
Duration of Overall Response (DOR) | 12 months
  Time from documentation of disease response to disease progression.
Progression-Free Survival (PFS) | 12 months
  PFS was defined as the time from CAR-T infusion to the date of disease progression or death from any cause. Participants not meeting the criteria for progression by the analysis data cutoff date were censored at their last evaluable disease assessment date.
Overall survival (OS) | 12 months
  OS was defined as the time from CAR-T infusion to the date of death. Participants who did not die by the analysis data cutoff date were censored at their last contact date.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiguo Long, Principal Investigator — Shanghai Pudong Hospital
Locations (1):
- Shanghai Pudong Hospital, Fudan University Affiliated Pudong Medical Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No